CLINICAL TRIAL: NCT02930733
Title: The Effects of Bilateral Serratus Plane Block on Postoperative Opioid Consumption After Breast Reduction Surgery
Brief Title: Serratus Plane Block For Breast Reduction Surgery
Acronym: SPB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, MD, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIA3
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Pain Management
Keywords: Postoperative Analgesia; Ultrasound guided serratus plane block
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ultrasound guided serratus plane block (Active Comparator): Bilateral ultrasound guided serratus plane block with 30 ml %0,25 bupivacaine
  Interventions: Drug: Bupivacaine
- ultrasound guided sham block (Placebo Comparator): Bilateral ultrasound guided sham block with 2 ml saline subcutaneously
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — 30 ml %0,25 bupivacaine bilaterally
  Arms: ultrasound guided serratus plane block
Drug: Saline — 2 ml saline subcutaneously bilaterally
  Arms: ultrasound guided sham block

SUMMARY:
Serratus plane block was first described in 2013 by Blanco and designed to primarily block the thoracic intercostal nerves. And this block provides sufficient analgesia lateral anterior and posterior part of thoracic wall.Increased use of ultrasound guidance for regional anesthesia in recent years has led to definition of thoracic wall PECs blocks by Blanco. The Serratus plain block (SPB), providing wider analgesia, with easier application and less adverse effects than neuroaxial blocks, has been defined after these blocks and has taken its place in the literature.In spite of the insufficient randomized clinical trials in the literature, SPB has been reported for many cases such as thoracoscopy, shoulder arthroscopy, breast surgery and axillary lymph node dissections, and the results are promising. The aim of this study is to determine effectiveness of ultrasound guided bilateral serratus plane block in patients undergoing breast reduction surgery.

Main outcome measures: The primary endpoint is postoperative opioid consumption.

Secondary endpoints are visual analogue pain scores, opioid related side effects.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients undergoing breast reduction surgery

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | First 24 hours total opioid consumption
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | postoperative first hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively.
Visual analog pain score | postoperative second hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at second hour postoperatively.
Visual analog pain score | postoperative 4th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 4th hour postoperatively.
Visual analog pain score | postoperative 8thhour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 8th hour postoperatively.
Visual analog pain score | postoperative 12th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 12th hour postoperatively.
Visual analog pain score | postoperative 24th hour
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at 24th hour postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ahiskalioglu, Principal Investigator — Ataturk University Anesthesiology and Reanimation
Locations (1):
- Ataturk University, Erzurum, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Background] Broseta AM, Errando C, De Andres J, Diaz-Cambronero O, Ortega-Monzo J. Serratus plane block: the regional analgesia technique for thoracoscopy? Anaesthesia. 2015 Nov;70(11):1329-30. doi: 10.1111/anae.13263. No abstract available. PMID 26449303